CLINICAL TRIAL: NCT02155387
Title: Extravascular Lung Water Index and Pulmonary Vascular Permeability Index Assessed by the Transpulmonary Thermodilution Method in Patients After Minimally Invasive Cardiac Surgery With Cardiopulmonary Bypass and One Lung Ventilation
Brief Title: Extravascular Lung Water and Pulmonary Vascular Permeability After Minimally Invasive Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Torsten Loop, M.D., Professor, University Hospital Freiburg
Other Study IDs: MICSLUWA2014
Record Dates: First submitted 2014-04-23; First posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: EVLW; EVLWI; PVPI; MICS
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Coronary artery bypass graft surgery: with cardiopulmonary bypass
- Pulmonary metastasectomy by thoracotomy: with one lung ventilation
- Minimal invasive mitral valve surgery: with cardiopulmonary bypass and one lung ventilation

SUMMARY:
The use of cardiopulmonary bypass (CPB) combined with one lung ventilation (OLV) allows to perform minimally invasive cardiac surgery (MICS) through small incisions. MICS is described to be associated with similar outcomes compared with conventional surgery. Although less invasive, MICS has not been reported to favorably impact the incidence of respiratory failure after surgery.

The combination CPB and OLV may induce acute respiratory distress syndrome (ARDS). After CPB contact of blood components with the artificial surface of the bypass, lung ischemia reperfusion injury (LIRI) and operative trauma may trigger a systemic inflammatory response syndrome (SIRS). During OLV, ARDS can result from hyperoxia, hyperperfusion and ventilatory distress in the ventilated lung as well as from LIRI and operative trauma of the collapsed lung.

Extravascular lung water (EVLW) includes all fluids in the lung except for those in the vascular compartment. An excess of EVLW may lead to respiratory insufficiency. This may be due to an increased hydrostatic intravascular pressure, as it occurs in cardiogenic pulmonary edema, and/or by an increase of lung endothelial and epithelial permeability, as in ARDS. The extravascular lung water index (EVLWI) assessed by the transpulmonary thermodilution technique may be a useful tool for accurate diagnosis of ARDS, and the pulmonary vascular permeability index (PVPI) may help in the differentiation between pulmonary edema due to an increase in the pulmonary capillary permeability versus an increase in the pulmonary capillary hydrostatic pressure.

As both CPB and OLV may induce an excess of EVLW, the investigators hypothesize that patients after MICS with intraoperative combination of CPB and OLV may have higher EVLWI and PVPI than those who received either CPB or OLV alone.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) occur with an incidence of 12% after cardiac surgery with the use of cardiopulmonary bypass (CBP). Using one-lung ventilation (OLV) in addition, as it is common practice in minimally invasive cardiac surgery (MICS), one can hypothesize that the risk for ARDS increases.

The objective of this prospective, observational study is to measure extravascular lung water index (EVLWI) and pulmonary vascular permeability index (PVPI) as parameters of lung edema through alteration in the pulmonary permeability by comparing three groups of surgery patients: I) patients with CPB, II) patients with OLV and III) patients with both CPB and OLV.

MICS allows coronary artery bypass grafting and cardiac valve surgery through small incisions, does not appear to be inferior to conventional surgery, but likely reduces postoperative pain, accelerates postoperative recovery and improves the cosmetic result. However, based on the available data, respiratory failure after MICS occurs at the same rate as after conventional cardiac surgery. In addition, unilateral re-expansion pulmonary edema, rarely seen after conventional cardiac surgery, has been described after MICS with CPB and OLV.

The pathophysiology of ARDS is characterized by massive inflammation that leads to a diffuse damage of both the alveolar epithelium and pulmonary vascular endothelium. Although the etiology of ARDS is multifactorial, the uniform result is an acute, nonhydrostatic, high-permeability lung injury with interstitial and alveolar protein-rich edema, epithelial damage and rapid onset of pulmonary fibrosis. This leads to the vast reduction of the pulmonary gas exchange and to hypoxemia.

Extravascular lung water (EVLW) comprises all fluids of the extravascular compartment of the lung, ie, intracellular water, lymphatic fluid, surfactant and extravasated plasma. Increased EVLW may be caused by an increased hydrostatic intravascular pressure, as it occurs in cardiogenic pulmonary edema, and/or by an increase of lung endothelial and epithelial permeability, as in ARDS. The EVLWI estimates the EVLW by using the transpulmonary thermodilution technique.The pulmonary vascular permeability index (PVPI) is the ratio between the EVLWI and the pulmonary blood volume, which is also measured by the transpulmonary thermodilution technique. The PVPI is thought to reflect the permeability of the alveolar-capillary barrier.

The combination of CPB and OLV permitted the development of MICS. CPB is an extracorporeal circulation, where a heart-lung machine takes over temporarily the pump function of the heart and the oxygenation and ventilation function of the lungs, thereby, allowing various heart and vascular surgical procedures. During CPB, blood from the right side of the heart is drained into the heart-lung machine and returned into the arterial system. This leads to a hypoperfusion of the lung, while blood flow is maintained only through the bronchial artery. OLV allows the surgeon to access the thorax cavity for the operation, while contralateral lung is ventilated.

It was originally thought that the lung is relatively resistant to ischemia due to its dual circulation. However, re-perfusion of the lung after CPB and/or OLV can trigger a fatal cascade, summarized as lung ischemia reperfusion injury (LIRI). LIRI involves intracellular injury and pertinent inflammatory responses, which result in apoptosis of the endothelium, alveolar capillary interstitial edema, hyaline membranization, and infiltration by neutrophils and macrophages. In addition, during CPB, the contact of blood components with the artificial surface of the bypass circuit contribute to the postoperative systemic inflammatory response syndrome (SIRS). Through these mechanisms, lung compliance and resistance as well as pulmonary permeability are affected, which contributes to the development of ARDS. During OLV, a combination of LIRI as well as surgical trauma and lung hyperinflation may lead to the release of inflammatory mediators which can alter endovascular permeability. Additionally, after thoracic surgery the pulmonary vascular permeability increases and re-expansion of the collapsed lungs may result in the so called re-expansion pulmonary edema.

To the best of the investigators knowledge, no study primarily aimed at examining the relationship between MICS and lung injury, although it is of high clinical interest whether the combination of CPB and OLV during MICS leads to increased EVLW and pulmonary permeability and ARDS.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years,
* written informed consent to participate in the study
* one of following surgeries: mitral valve surgery with CPB, resection of pulmonary metastases with OLV, or minimally invasive mitral valve surgery with CPB and OLV.

Exclusion Criteria:

* chronic respiratory insufficiency
* history of pulmonary resection or pneumonectomy
* pulmonary thromboembolism
* lung injury
* severe peripheral arterial disease
* emergency surgery
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 18 and 75 years who need one of following surgeries: coronary artery bypass graft surgery with CPB, resection of pulmonary metastases with OLV, or minimally invasive mitral valve surgery with CPB and OLV.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Extravascular lung water index (EVLWI) measured by a Pulse Contour Cardiac Output (PiCCO©) system device | T0= baseline; Ta= 15 minutes after start of the OLV; Tb=15 minutes after stop of the CPB while still under OLV; 30 minutes (T1), 6 hours (T2), 12 hours (T3) and 24 hours (T4) after stop of OLV and/or CPB.
  EVLWI (ml/Kg) will be assessed after the induction of general anesthesia but before the surgery starts. This observational point is defined as T0. The observational time points T1, T2, T3 and T4 are 30 minutes, 6 hours, 12 hours and 24 hours, respectively, after stop of OLV and/or CPB. In case of OLV, an observational time point (Ta) will be added 15 minutes after start of the OLV. In patients with CPB and OLV, an additional time point (Tb) is 15 minutes after stop of the CPB while still under OLV.
Pulmonary vascular permeability index (PVPI) measured by a Pulse Contour Cardiac Output (PiCCO©) system device | T0, T1, T2, T3, T4, Ta, Tb
  PVPI will be assessed after the induction of general anesthesia but before the surgery starts. This observational point is defined as T0. The observational time points T1, T2, T3 and T4 are 30 minutes, 6 hours, 12 hours and 24 hours, respectively, after stop of OLV and/or CPB. In case of OLV, an observational time point (Ta) will be added 15 minutes after start of the OLV. In patients with CPB and OLV, an additional time point (Tb) is 15 minutes after stop of the CPB while still under OLV.

SECONDARY OUTCOMES:
Any respiratory problem that the patient had during the postoperative period in the intensive care unit | one month after the surgery
  One month after the surgery, any respiratory problem, such as infiltrate, atelectasis, pleural fluid, pneumonia or ARDS, that the patient had during the postoperative recovery period in the intensive care unit (ICU) will be assessed based on the medical records. Chest radiograph will be reviewed to assess the presence of infiltrates, atelectasis, pleural fluid and pulmonary edema. The pneumonia diagnosis will be based on the presence of pulmonary infiltrates and laboratory results. The Berlin definition will be used to establish the diagnosis of ARDS.

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Loop, MD,Professor, Principal Investigator — University Hospital Freiburg
Locations (1):
- Departement of Anaesthesiology and Critical Care Medicine, University Medical Center, Freiburg im Breisgau, Baden-Wurttemberg, Germany